CLINICAL TRIAL: NCT01810120
Title: Phase I/II Study of Allogeneic Hematopoietic Stem Cell Transplantation From an HLA-partially Matched Family Donor After TCR Alfa Beta Negative Selection in Pediatric Patients Affected by Hematological Disorders
Brief Title: Trial to Assess the Efficacy of a TCR Alfa Beta Depleted Graft in Pediatric Affected by ALL or AML and Receiving an HSCT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mariella Enoc (Other)
Responsible Party: Sponsor-Investigator, Mariella Enoc, Director Department of Pediatric Hematology and Oncology, Bambino Gesù Hospital and Research Institute
Organization: Bambino Gesù Hospital and Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OPBG_359.11
Record Dates: First submitted 2012-01-17; First posted 2013-03-13 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Acute Lymphoblastic Leukemia; Leukemia Acute Myeloid - AML; Non-Hodgkin Lymphoma; Myelodysplastic Syndromes
Keywords: Hematologic; Malignant; Non-Malignant; Allogeneic; Transplant; Non-Hodgkin Lymphoma; Pediatric; Acute lymphoblastic leukemia; Acute Myeloid leukemia; Myelodysplastic Syndromes; T cells receptor alfa beta
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Non-Hodgkin; Myelodysplastic Syndromes; Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TCR alfa beta depleted graft, infusion (Experimental): The leukapheresis product will undergo TCR alfa beta negative selection following the standardized protocol.
  Interventions: Biological: TCR alfa beta T cell depletion

INTERVENTIONS:
Biological: TCR alfa beta T cell depletion — total nucleated cells from the leukapheresis product will undergo TCR alfa beta negative selection and the product of the depletion will be infused to the patient
  Other Names: nucleated cells

SUMMARY:
Allocation: Non-Randomized Endpoint Classification: Safety/Feasibility Intervention Model: Single Group Assignment Masking: Open Label Primary Purpose: Treatment Study to assess the feasibility and safety of the infusion of a T cells receptor (TCR) alfa beta depleted graft in pediatric patients affected by malignant and non-malignant hematological disorders and receiving an Hematopoietic stem cell transplantation (HSCT) from a Human leukocyte antigen (HLA) partially matched family donor.

DETAILED DESCRIPTION:
In this study the hypothesis is that the transplantation of Peripheral blood stem cells (PBSC)selectively depleted of TCR alfa beta T lymphocytes would offers some advantages over the use of positively selected CD34+ stem cells because of the presence of other non-stem ancillary cells (in particular Natural killer (NK) and alfa beta T cells) that might have potential positive effects on the outcome of the transplant.

The clinical relevance of NK-cell alloreactivity has been demonstrated in adult patients affected by Acute myeloid leukemia (AML) and given T-cell depleted HSCT from an HLA-disparate relative where a subgroup of patients had a particularly low risk of leukemia relapse. These patients belonged to the group transplanted from a donor having NK cells that were alloreactive towards recipient targets i.e. the patient cells express HLA-class I alleles that do not share the inhibiting allelic determinants recognized by Killer immunoglobulin-like receptors (KIR) on donor NK cells. The emergence of this concept of NK-cell alloreactivity has represented a sort of revolution in the field of Haplo-identical hematopoietic stem cell translantation (haplo-HSCT), as the presence of alloreactive NK cells has been shown to positively affect the outcome of transplantation in adults and to display a Graft versus leukemia (GvL) effect that can compensate for the lack of T-specific anti-tumor effect.

The purpose of this study is to evaluate the feasibility and safety of the selective infusion of TCR alfa beta T cell depleted graft in pediatric patients affected by malignant or non malignant hematological disorders and receiving an HSCT from a partially matched family donor.

This study will provide new data on the feasibility and the safety of using a TCR alfa beta T cell depleted graft instead of fully T cell depleted graft to improve the outcome of patients receiving a haplo-HSCT for the treatment of hematological disorders.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 3 months and < 21 years
* Patients diagnosed with malignant hemopathies (Acute Lymphoblastic leukemia (ALL), Acute Myeloid Leukemia (AML), Non-Hodgkin Lymphoma (NHL)) in complete morphological remission or Myelodysplastic Syndromes (MDS), Solid Tumors or non malignant hematological disorders (SCID, Acquired and Congenital Aplastic Anemia, other Primary Immunodeficiencies, Life-threatening Cytopenia) eligible for an allogeneic transplantation and lacking a related or unrelated HLA-matched donor
* Patients displaying an HLA-partially matched family donor
* Lansky/Karnofsky score > 40, WHO > 4
* Signed written informed consent

Exclusion Criteria:

* Grade >II acute GvHD or chronic extensive GvHD at the time of inclusion
* Patient receiving an immunosuppressive treatment for GvHD treatment at the time of inclusion
* Dysfunction of liver (ALT/AST > 5 times normal value, or bilirubin > 3 times normal value), or of renal function (creatinine clearance < 30 ml / min)
* Severe cardiovascular disease (arrhythmias requiring chronic treatment, congestive heart failure or left ventricular ejection fraction <40%)
* Current active infectious disease (including positive HIV serology or viral RNA)
* Serious concurrent uncontrolled medical disorder
* Pregnant or breast feeding female patient
* Lack of parents' informed consent.

Ages: 3 Months to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
CD34+ cells | up to 3 month
  Target number of CD34+ cells in at least 80% of the patients

SECONDARY OUTCOMES:
Primary and secondary graft failure | up to 24 months after transplantation
  Cumulative incidence of primary and secondary graft failure
Acute and chronic GvHD | up to 24 months after transplantation
  Cumulative incidence and severity of acute and chronic GvHD occurring after the transplantation
Overall survival (OS) and disease-free survival | up to 24 months after transplantation
  The overall survival (OS) and disease-free survival probability compared with a cohort of historical controls
TCR alfa beta cells | up to 12 months after the transplantation
  The immunological reconstitution of TCR alfa beta cells compared with a cohort of historical controls

CONTACTS AND LOCATIONS:
Overall Officials: Franco Locatelli, Prof, Principal Investigator — Bambino Gesù Children's Hospital
Locations (1):
- Department of Oncology/Hematology of the Hospital Bambino Gesù (Roma), Rome, Italy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Copelan EA. Hematopoietic stem-cell transplantation. N Engl J Med. 2006 Apr 27;354(17):1813-26. doi: 10.1056/NEJMra052638. No abstract available. PMID 16641398
- [Background] Rocha V, Locatelli F. Searching for alternative hematopoietic stem cell donors for pediatric patients. Bone Marrow Transplant. 2008 Jan;41(2):207-14. doi: 10.1038/sj.bmt.1705963. Epub 2007 Dec 17. PMID 18084331
- [Background] Gluckman E. Cord blood transplantation. Biol Blood Marrow Transplant. 2006 Aug;12(8):808-12. doi: 10.1016/j.bbmt.2006.05.011. No abstract available. PMID 16864050
- [Background] Locatelli F, Pende D, Maccario R, Mingari MC, Moretta A, Moretta L. Haploidentical hemopoietic stem cell transplantation for the treatment of high-risk leukemias: how NK cells make the difference. Clin Immunol. 2009 Nov;133(2):171-8. doi: 10.1016/j.clim.2009.04.009. Epub 2009 May 29. PMID 19481979
- [Background] Martelli MF, Aversa F, Bachar-Lustig E, Velardi A, Reich-Zelicher S, Tabilio A, Gur H, Reisner Y. Transplants across human leukocyte antigen barriers. Semin Hematol. 2002 Jan;39(1):48-56. doi: 10.1053/shem.2002.29255. PMID 11799529
- [Background] Reisner Y, Kapoor N, Kirkpatrick D, Pollack MS, Cunningham-Rundles S, Dupont B, Hodes MZ, Good RA, O'Reilly RJ. Transplantation for severe combined immunodeficiency with HLA-A,B,D,DR incompatible parental marrow cells fractionated by soybean agglutinin and sheep red blood cells. Blood. 1983 Feb;61(2):341-8. PMID 6217853
- [Background] Antoine C, Muller S, Cant A, Cavazzana-Calvo M, Veys P, Vossen J, Fasth A, Heilmann C, Wulffraat N, Seger R, Blanche S, Friedrich W, Abinun M, Davies G, Bredius R, Schulz A, Landais P, Fischer A; European Group for Blood and Marrow Transplantation; European Society for Immunodeficiency. Long-term survival and transplantation of haemopoietic stem cells for immunodeficiencies: report of the European experience 1968-99. Lancet. 2003 Feb 15;361(9357):553-60. doi: 10.1016/s0140-6736(03)12513-5. PMID 12598139
- [Background] Bachar-Lustig E, Rachamim N, Li HW, Lan F, Reisner Y. Megadose of T cell-depleted bone marrow overcomes MHC barriers in sublethally irradiated mice. Nat Med. 1995 Dec;1(12):1268-73. doi: 10.1038/nm1295-1268. PMID 7489407
- [Background] Reisner Y, Martelli MF. Stem cell escalation enables HLA-disparate haematopoietic transplants in leukaemia patients. Immunol Today. 1999 Aug;20(8):343-7. doi: 10.1016/s0167-5699(98)01428-5. PMID 10431152
- [Background] Aversa F, Tabilio A, Terenzi A, Velardi A, Falzetti F, Giannoni C, Iacucci R, Zei T, Martelli MP, Gambelunghe C, et al. Successful engraftment of T-cell-depleted haploidentical "three-loci" incompatible transplants in leukemia patients by addition of recombinant human granulocyte colony-stimulating factor-mobilized peripheral blood progenitor cells to bone marrow inoculum. Blood. 1994 Dec 1;84(11):3948-55. PMID 7524753
- [Background] Aversa F, Tabilio A, Velardi A, Cunningham I, Terenzi A, Falzetti F, Ruggeri L, Barbabietola G, Aristei C, Latini P, Reisner Y, Martelli MF. Treatment of high-risk acute leukemia with T-cell-depleted stem cells from related donors with one fully mismatched HLA haplotype. N Engl J Med. 1998 Oct 22;339(17):1186-93. doi: 10.1056/NEJM199810223391702. PMID 9780338
- [Background] Aversa F, Terenzi A, Tabilio A, Falzetti F, Carotti A, Ballanti S, Felicini R, Falcinelli F, Velardi A, Ruggeri L, Aloisi T, Saab JP, Santucci A, Perruccio K, Martelli MP, Mecucci C, Reisner Y, Martelli MF. Full haplotype-mismatched hematopoietic stem-cell transplantation: a phase II study in patients with acute leukemia at high risk of relapse. J Clin Oncol. 2005 May 20;23(15):3447-54. doi: 10.1200/JCO.2005.09.117. Epub 2005 Mar 7. PMID 15753458
- [Background] Ciceri F, Labopin M, Aversa F, Rowe JM, Bunjes D, Lewalle P, Nagler A, Di Bartolomeo P, Lacerda JF, Lupo Stanghellini MT, Polge E, Frassoni F, Martelli MF, Rocha V; Acute Leukemia Working Party (ALWP) of European Blood and Marrow Transplant (EBMT) Group. A survey of fully haploidentical hematopoietic stem cell transplantation in adults with high-risk acute leukemia: a risk factor analysis of outcomes for patients in remission at transplantation. Blood. 2008 Nov 1;112(9):3574-81. doi: 10.1182/blood-2008-02-140095. Epub 2008 Jul 7. PMID 18606875
- [Background] Klingebiel T, Cornish J, Labopin M, Locatelli F, Darbyshire P, Handgretinger R, Balduzzi A, Owoc-Lempach J, Fagioli F, Or R, Peters C, Aversa F, Polge E, Dini G, Rocha V; Pediatric Diseases and Acute Leukemia Working Parties of the European Group for Blood and Marrow Transplantation (EBMT). Results and factors influencing outcome after fully haploidentical hematopoietic stem cell transplantation in children with very high-risk acute lymphoblastic leukemia: impact of center size: an analysis on behalf of the Acute Leukemia and Pediatric Disease Working Parties of the European Blood and Marrow Transplant group. Blood. 2010 Apr 29;115(17):3437-46. doi: 10.1182/blood-2009-03-207001. Epub 2009 Dec 29. PMID 20040760
- [Background] Trinchieri G. Biology of natural killer cells. Adv Immunol. 1989;47:187-376. doi: 10.1016/s0065-2776(08)60664-1. PMID 2683611
- [Background] Moretta L, Ciccone E, Mingari MC, Biassoni R, Moretta A. Human natural killer cells: origin, clonality, specificity, and receptors. Adv Immunol. 1994;55:341-80. doi: 10.1016/s0065-2776(08)60513-1. No abstract available. PMID 7508176
- [Background] Moretta L, Moretta A. Unravelling natural killer cell function: triggering and inhibitory human NK receptors. EMBO J. 2004 Jan 28;23(2):255-9. doi: 10.1038/sj.emboj.7600019. Epub 2003 Dec 18. PMID 14685277
- [Background] Moretta A, Bottino C, Mingari MC, Biassoni R, Moretta L. What is a natural killer cell? Nat Immunol. 2002 Jan;3(1):6-8. doi: 10.1038/ni0102-6. No abstract available. PMID 11753399
- [Background] Moretta A, Locatelli F, Moretta L. Human NK cells: from HLA class I-specific killer Ig-like receptors to the therapy of acute leukemias. Immunol Rev. 2008 Aug;224:58-69. doi: 10.1111/j.1600-065X.2008.00651.x. PMID 18759920
- [Background] Janeway CA Jr, Medzhitov R. Innate immune recognition. Annu Rev Immunol. 2002;20:197-216. doi: 10.1146/annurev.immunol.20.083001.084359. Epub 2001 Oct 4. PMID 11861602
- [Background] Parham P. Innate immunity: The unsung heroes. Nature. 2003 May 1;423(6935):20. doi: 10.1038/423020a. No abstract available. PMID 12721604
- [Background] Pende D, Marcenaro S, Falco M, Martini S, Bernardo ME, Montagna D, Romeo E, Cognet C, Martinetti M, Maccario R, Mingari MC, Vivier E, Moretta L, Locatelli F, Moretta A. Anti-leukemia activity of alloreactive NK cells in KIR ligand-mismatched haploidentical HSCT for pediatric patients: evaluation of the functional role of activating KIR and redefinition of inhibitory KIR specificity. Blood. 2009 Mar 26;113(13):3119-29. doi: 10.1182/blood-2008-06-164103. Epub 2008 Oct 22. PMID 18945967
- [Background] Hayday AC. Gammadelta T cells and the lymphoid stress-surveillance response. Immunity. 2009 Aug 21;31(2):184-96. doi: 10.1016/j.immuni.2009.08.006. PMID 19699170
- [Derived] Merli P, Algeri M, Galaverna F, Bertaina V, Lucarelli B, Boccieri E, Becilli M, Quagliarella F, Rosignoli C, Biagini S, Girolami E, Meschini A, Del Principe G, Sborgia R, Catanoso ML, Carta R, Strocchio L, Pinto RM, Buldini B, Falco M, Meazza R, Pende D, Andreani M, Li Pira G, Pagliara D, Locatelli F. TCRalphabeta/CD19 cell-depleted HLA-haploidentical transplantation to treat pediatric acute leukemia: updated final analysis. Blood. 2024 Jan 18;143(3):279-289. doi: 10.1182/blood.2023021336. PMID 37738655
- [Derived] Merli P, Pagliara D, Galaverna F, Li Pira G, Andreani M, Leone G, Amodio D, Pinto RM, Bertaina A, Bertaina V, Mastronuzzi A, Strocchio L, Boccieri E, Pende D, Falco M, Di Nardo M, Del Bufalo F, Algeri M, Locatelli F. TCRalphabeta/CD19 depleted HSCT from an HLA-haploidentical relative to treat children with different nonmalignant disorders. Blood Adv. 2022 Jan 11;6(1):281-292. doi: 10.1182/bloodadvances.2021005628. PMID 34592755
- [Derived] Strocchio L, Pagliara D, Algeri M, Li Pira G, Rossi F, Bertaina V, Leone G, Pinto RM, Andreani M, Agolini E, Girardi K, Gaspari S, Grapulin L, Del Bufalo F, Novelli A, Merli P, Locatelli F. HLA-haploidentical TCRalphabeta+/CD19+-depleted stem cell transplantation in children and young adults with Fanconi anemia. Blood Adv. 2021 Mar 9;5(5):1333-1339. doi: 10.1182/bloodadvances.2020003707. PMID 33656536
- [Derived] Locatelli F, Merli P, Pagliara D, Li Pira G, Falco M, Pende D, Rondelli R, Lucarelli B, Brescia LP, Masetti R, Milano GM, Bertaina V, Algeri M, Pinto RM, Strocchio L, Meazza R, Grapulin L, Handgretinger R, Moretta A, Bertaina A, Moretta L. Outcome of children with acute leukemia given HLA-haploidentical HSCT after alphabeta T-cell and B-cell depletion. Blood. 2017 Aug 3;130(5):677-685. doi: 10.1182/blood-2017-04-779769. Epub 2017 Jun 6. PMID 28588018
- [Derived] Airoldi I, Bertaina A, Prigione I, Zorzoli A, Pagliara D, Cocco C, Meazza R, Loiacono F, Lucarelli B, Bernardo ME, Barbarito G, Pende D, Moretta A, Pistoia V, Moretta L, Locatelli F. gammadelta T-cell reconstitution after HLA-haploidentical hematopoietic transplantation depleted of TCR-alphabeta+/CD19+ lymphocytes. Blood. 2015 Apr 9;125(15):2349-58. doi: 10.1182/blood-2014-09-599423. Epub 2015 Jan 22. PMID 25612623
- [Derived] Bertaina A, Merli P, Rutella S, Pagliara D, Bernardo ME, Masetti R, Pende D, Falco M, Handgretinger R, Moretta F, Lucarelli B, Brescia LP, Li Pira G, Testi M, Cancrini C, Kabbara N, Carsetti R, Finocchi A, Moretta A, Moretta L, Locatelli F. HLA-haploidentical stem cell transplantation after removal of alphabeta+ T and B cells in children with nonmalignant disorders. Blood. 2014 Jul 31;124(5):822-6. doi: 10.1182/blood-2014-03-563817. Epub 2014 May 28. PMID 24869942